CLINICAL TRIAL: NCT01874639
Title: Use of Transcollation Device to Decrease Blood Loss During Hepatic Resections: a Randomized Cohort Study
Brief Title: Use of Transcollation Device to Decrease Blood Loss During Hepatic Resections: a Randomized Cohort Study (HEPACOLL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: INNOPATH (Unknown); MEDTRONIC labs provide the aquamantys® probes for the study. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-0156
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Hepatectomy
Keywords: Hepatectomy; blood loss; hemostasis; coagulation; Liver surgery (benign or malign); Resection of 2 or more segments
MeSH Terms: conditions — Hemorrhage; Thrombosis

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- hepatectomy ( conventional hemostasis ) (Experimental): After validation of the inclusion and exclusion criteria, the patients include in this clinical trial will be randomized between the two arms of the study:
  - Control group: hepatectomy with conventional hemostasis using standard bipolar coagulation
  Interventions: Device: standard bipolar coagulation
- hepatectomy with Aquamantys (Other): After validation of the inclusion and exclusion criteria, the patients include in this clinical trial will be randomized between the two arms of the study:
  - Test group: hepatectomy with Aquamantys®
  Interventions: Device: Aquamantys® probe for liver hemostasis

INTERVENTIONS:
Device: standard bipolar coagulation
  Arms: hepatectomy ( conventional hemostasis )
Device: Aquamantys® probe for liver hemostasis
  Arms: hepatectomy with Aquamantys

SUMMARY:
Blood loss in hepatic surgery is the main factor of postoperative morbidity. The use of the most effective possible tool for hemostasis allows a bleeding decrease during liver transection and thus could reduce postoperative morbidity.

In the past decade, the improvement of techniques of transection of the hepatic parenchyma was one of the most important factors to ensure the hepatectomy safety. But the clinical performances of these technological innovations (ultrasound dissectors, monopolar radiofrequency probes and dissection devices using pressurized water) remain still unclear.

The medical device of hemostasis Aquamantys® (Salient company, Innopath) use the technology of "transcollation" combining a source of radiofrequency associated with a conductive liquid (NaCl 0.9% solution). The system consists of a specific generator (Aquamantys Pump Generator®) and single-use probes (Aquamantys 2.3 BipolarSealer®). The energy of radiofrequency is delivered by two bipolar electrodes. The innovative aspect of this device consists in maintaining the tissue to a temperature of 100°C, while using a conductive liquid which acts as process of cooling and avoids the drying out of tissues, smoke, risks of electric arc and overheating met with conventional electrosurgery. This device allows the coagulation of blood vessels but also bile ducts. The Aquamantys® system could decrease the postoperative morbidity and mortality due to a decrease of blood loss and biliary leak. These clinical benefits could be translated by an improvement of the direct and indirect costs associated to the surgery. However the Aquamantys® technology has not been scientifically validated in the context of the hepatic surgery, and this technology is expensive due to the purchase of single-use bipolar probes (Aquamantys 2.3 BipolarSealer®) and to the investment in a generator (Aquamantys Pump Generator®).

Consequently, it is essential to realize a study measuring the clinical and medical economic impact of the transcollation technology (Aquamantys® device) in the hepatic surgery.

DETAILED DESCRIPTION:
After validation of the inclusion and exclusion criteria, the patients include in this clinical trial will be randomized between the two arms of the study:

* Control group: hepatectomy with conventional hemostasis using standard bipolar coagulation
* Test group: hepatectomy with Aquamantys®

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery for liver resection of malignant or benign disease
* Hepatic resection of two or more segments
* No coagulation disorder
* No portal hypertension (platelets ≥ 100 G/L, absence of splenomegaly, absence of portal hypertension varices)
* Obtaining the patient's written consent

Exclusion Criteria:

* Age < 18 years and > 80 years
* ASA score > 3
* Cirrhosis, liver fibrosis > F2, steatosis > 60%, sinusoidal obstruction syndrome
* Cognitive troubles and major disability making impossible to understand the study and signed the informed consent (e.g. dementia, psychiatric disorders like psychosis, speech disorder ...)
* Liver and kidney failure
* Pregnancy and lactating women
* Legal incapacity
* Patients already enrolled in a clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Blood loss during surgery | at day 0

SECONDARY OUTCOMES:
Duration of liver transection | at day 0
Duration of surgery | at day 0
Duration of hospital stay | at day 1
Number of red blood cells transfusions | at day 0
Number of frozen plasma transfusions | at day 0
Volume of crystalloid and colloid fluids | at day 0
Need of norepinephrine during the surgery | at day 0

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel BUC, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France